CLINICAL TRIAL: NCT07365865
Title: Dimensional Changes of the Keratinized Mucosa in Edentulous Ridges Following Accordian Technique Versus Conventional Free Gingival Grafts: A Randomized Clinical Trial
Brief Title: Dimensional Changes of the Keratinized Mucosa in Edentulous Ridges Following Accordian Technique Versus Conventional Free Gingival Grafts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Essam Mohamed Khalifa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FGG by Accordian technique
Record Dates: First submitted 2025-09-30; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Deficient Keratinized Mucosa; Healthy
Keywords: free gingival graft; Accordian; keratinized mucosa

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group ( Accordian Group ) (Experimental): steps from 1-7 as Active comparator group + 7 -Free gingival graft will be harvested from the palatal area, as previously mentioned, with a length of 40% of the mesiodistal length of the recipient area. Intermittent incisions to cover the whole length of the recipient area. 8- The graft will be located at the recipient area, and sutured with interrupted sutures.
  Interventions: Procedure: Expanded mesh free gingival graft ( Accordian technique )
- Conventional free gingival graft (Active Comparator): 1- Infiltration anesthesia at the recipient area. 2- A horizontal incision, 0.5mm above the mucogingival junction extending along the area of the missing teeth. 3-Two vertical incisions diverging slightly in a corono-apical direction and extending into the alveolar mucosa. 4-The trapezoidal area will be dissected split thickness to expose the periosteum. 5-Infiltration anesthesia at the palatal area. 6-The free gingival graft will be harvested from the palate consisting of epithelial connective tissue of thickness more than 1mm.7- The palatal graft thickness will be determined by the coronal horizontal incision and the releasing incisions. The blade will be inserted perpendicular to the underlying deep tissue layers to a depth equal to the required graft thickness. 8- The graft will be harvested by inclining the blade horizontally, keeping it parallel to the external mucosal plane.9- The graft will be located at the recipient area, and sutured with interrupted sutures.
  Interventions: Procedure: conventional free gingival graft

INTERVENTIONS:
Procedure: Expanded mesh free gingival graft ( Accordian technique ) — Free gingival graft by expanded free gingival graft
  Arms: Interventional group ( Accordian Group )
Procedure: conventional free gingival graft — conventional free gingival graft
  Arms: Conventional free gingival graft

SUMMARY:
Inadequacy of the attached keratinized tissue (<2 mm) affects the long-term maintenance of prostheses and implants due to poor oral hygiene, plaque accumulation, inflammation, bleeding on probing, gingival recession , attachment loss, and crestal bone loss .Consequently, keratinized tissue augmentation is considered to compensate for keratinized attached gingival width inadequacy. Lack of keratinized tissue (KT) or KT with a narrow width (≤2 mm) compromise the long-term maintenance of peri-implant tissue health . Peri-implantitis was more frequently detected at dental implants sites with reduced width of KT than at those with adequate KT width.

Free gingival graft (FGG) is regarded as an efficient method with significant clinical application . However, following harvesting larger grafts, some limitations arise in the donor site. Extensive palatal wound may cause discomfort and morbidity for the patient, the rugae area is unsuitable for graft material and the greater palatine artery will be of a great concern.

DETAILED DESCRIPTION:
Free gingival graft with accordion technique can expand the tissue up to 50%, and cover the recipient bed 1.5 times longer than the original graft by its alternating incisions on both edges. This avoids high rate of complications and limited amount of palatal mucosa available for grafting. It allows for the harvesting of smaller size, reducing patient morbidity and post-operative pain for augmenting wide areas. The area between the alternate incisions become epithelized with keratinized tissue by creeping of the surrounding tissues . Also, it provides having proper keratinized tissue width at large edentulous areas.

An adequate amount of keratinized tissue is required to maintain periodontal health and gingival recession . In order to preserve gingival health, a 2mm of keratinized gingiva is required. Keratinized tissue width is considered insufficient around teeth if it is below 2mm, where it will be associated with less vertical dimension, uncomfortable brushing, and unfavorable peri-implant conditions. Moreover, it was proven to be a risk factor for the severity of the peri-implant mucositis.

Wide zone of keratinized mucosa has a role in preservation of soft and hard tissue stability around dental implants, and with their long-term maintenance . Thick soft tissues have a positive impact on mucosal margin stability by reducing the mid-buccal soft tissue recession. Dental implants with lower KT width (<2 mm) were more likely to have peri-implantitis than those with adequate KT width (≥2 mm). Moreover, they are associated with higher plaque and bleeding scores .

Soft tissue augmentation is considered to increase the soft tissue volume as well as the keratinized mucosa. These plastic procedures re-establish the functional and biological stability , cleansibilty of the prosthesis and aesthetics . Soft tissue augmentation can be performed prior to implant placement, simultaneously with second stage surgery or after insertion of the final prosthesis.

The free gingival graft (FGG) and the subepithelial connective tissue graft (SCTG) are from the autogenous soft tissue grafting procedures used for the augmentation of keratinized tissue . Free gingival graft is indicated to increase the attached gingiva, elimination of the frenum and muscular attachments, root coverage, and vestibular extension.

The main disadvantage of the autogenous tissue grafts is that the harvesting procedure leads to prolonged healing at the donor site and patient's morbidity . The amount of soft-tissue that can be harvested form the palatal mucosa is often limited thus covering broad mucosal areas can be a real challenge. Also, the hard palate has anatomical limitation of the greater palatine artery at the posterior palate and at the front of the rugae . Patients frequently express discomfort and paresthesia for a few weeks following surgery.

In the augmentation of wide area, we encounter limitations in the autogenous donor tissue, so many grafting modifications have been suggested in an effort to reduce the requirement for a large autograft harvest. In the accordion technique, which was introduced by Rateitschak et al. in 1985, the FGG was enlarged, by making alternating incisions with a scalpel blade at different sides of the graft. Allowing to expand the tissue up to nearly 50%. The strip gingival autograft technique was first described by Han in 1983. In this approach, thin strips of FGGs were positioned parallel to one another and secured to the prepared periosteal bed's most apical extension, allowing the exposed connective tissue area in between the graft strips to mend secondary intention .

In 2004, Akbari proposed a vertical modification of the strip gingival graft. Another modification by Urban et al. by combining the strip gingival graft technique with the xenogeneic collagen matrix (CM) to address the extensive areas of mucogingival alterations resulting from advanced regenerative procedures. One of the most effective techniques for soft tissue augmentation is the apically positioned flap in conjunction with the free gingival graft, even if alternative therapies such as apically positioned flap alone, collagen matrix, and acellular dermal matrix have been developed A recent systematic review and meta-analyses assessed the effectiveness of several surgical techniques intended to restore the adequate level of keratinized mucosa at implant locations . The best method for increasing the amount of keratinized tissue surrounding dental implants is the free gingival graft. When allograft was utilized rather of xenograft, comparable results were documented .

To overcome the limitation of the donor site in the conventional FGG, Rateitschak et al. proposed to modify the harvested graft extra-orally aiming to expand its size by making alternate incisons by 50%, allowing harvesting tissue with smaller size. Consequently, reducing patient morbidity, which is considered the main advantage of the accordion technique. In the healing phase, keratinized tissue from the neighboring area creeps in and epithelializes the spaces between the wounds. This creeping process is not always predictable. One of this method's drawback is the lack of a defined standard for the intervals between incisions that keratinized epithelium from the creeping process can cover. Shrinkage is a normal process following FGG treatment, in contrast to the creeping process.

Correspondingly, this tissue expanding leads to harvesting less tissue and subsequently decreased pain and morbidity. Dimensional changes of the grafted tissue cause not to remain the initial amount of the keratinized mucosa. Studies have documented a wide spectrum of shrinkage, primarily associated with the traditional technique. Therefore, considering the limitations in donor tissue, the accordion technique is a suitable option. However, because there is no set standard for incisions and there may be some creeping and shrinkage involved, conventional and accordion FGG were to be compared for changes in vertical dimensions and clinical outcomes.

One of the main concerns after grafting is shrinkage of the graft, which occurs due to muscle repositioning and muscle contraction after one month from the surgery. The majority of the investigations have focused on the dimensional changes of FGG around teeth with limited evidence in edentulous ridges.

Based on the previous studies, dimensional changes occur after soft tissue augmentation by free gingival graft. Thus, the current trial is conducted to evaluate dimensional changes occurs following conventional free gingival graft and free gingival graft by accordion technique in edentulous ridges prior to implant placement, to reduce patient pain and morbidity in large areas, as well as provide adequate keratinized attached gingiva for the future restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with apico-coronal keratinized tissue width less than 2 millimeters
* Edentulous area with at least 2 missing teeth
* No systemic disease or active periodontitis
* Non smoker
* Age ≥ 20 years old .
* Plaque index and bleeding index < 25%.
* Teeth loss with medium to thick gingival biotype (Periodontal probe not visible when inserted into the buccal gingival margin).
* Fully autonomous behavior and expression ability with good compliance.

Exclusion Criteria:

* Patients with any systemic disease
* Patients with symptoms such as inflammation, bleeding on probing, or pus discharge.
* Poor oral hygiene
* Adjacent teeth with acute and chronic tooth disease at the implant site
* Smokers ≥ 10 cigarettes/day.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Vertical graft shrinkage % | Baseline 3 months
  Vertical graft shrinkage will be measured using UNC 15 Periodontal probe from reference point that will be taken (mid of the ridge) from where the graft will be sutured 3 months post-surgery

SECONDARY OUTCOMES:
Apico coronal keratinized tissue width | Baseline 3 months
  Changes in keratinized tissue width will be measured with UNC 15 Periodontal probe by roll test from reference point that will be taken (mid of the ridge) from where the graft will be sutured 3 after surgery
Vestibular depth | Baseline 3 months
  Vestibular depth will be measured from reference point that will be taken (mid of the ridge) from where the graft will be sutured to the greatest concavity of the mucobuccal fold by UNC 15 periodontal probe 3 post-surgery
Keratinized tissue thickness | Baseline 3 months
  Keratinized tissue thickness will be measured through transgingival probing by applying local anesthesia and using UNC 15 periodontal probe with a silicone stopper to be inserted perpendicular in the soft tissue until feeling resistance (Hitting buccal bone), at 1, 3 and 5 mm beyond the midcrest of the ridge. Then the distance between the silicone stopper and the tip of the probe will be measured 3 and 6 months after surgery
Post surgical pain assessment | Day 1 Day 3 Day 14
  Readings will be recorded by the patient on the day of surgery, on the next two days after surgery and on the day of suture removal using the VAS which is a descriptive numerical rating scale of 0 to 10 0= No pain 1-3= Mild pain 4-6= Moderate pain 7-10= Severe pain
Patient satisfaction | 3 months
  A 2-item questionnaire will be given to the patients to be answered using a 7-point answer scale for assessing their satisfaction for the whole procedure and results obtained.
  0 is the minimum satisfaction 7 is the maximum satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo university, Cairo, Egypt